CLINICAL TRIAL: NCT03798431
Title: MINDFUL-OBOT Pilot: Effect of Mindfulness on Opioid Use and Anxiety During Primary Care Buprenorphine Treatment -- Pilot Study
Brief Title: MINDFUL-OBOT: Effect of Mindfulness on Opioid Use and Anxiety During Primary Care Buprenorphine Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-1094/08/18; R21AT010125 (NIH)
Record Dates: First submitted 2018-12-10; First posted 2019-01-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder; Anxiety; Depression; Stress Related Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: There will be no randomization for this pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- M-ROCC (Experimental): Mindful Recovery OUD Care Continuum (M-ROCC) builds on other mindfulness interventions for addictive disorders, but is specifically designed with the clinical needs of OUD patients on buprenorphine and logistic needs of primary care OBOT clinicians in mind. It focuses on integration of mindfulness practice for living well through stress, anxiety, depression, pain and addiction recovery. M-ROCC curriculum has three primary components, including a low-dose mindfulness phase, an intensive mindfulness training phase and then ongoing mindful recovery support.
  Interventions: Behavioral: M-ROCC

INTERVENTIONS:
Behavioral: M-ROCC — 1. LDM (Low-Dose Mindfulness): A 4-wk intro mindfulness program for OUD, 50 min/week including explicit training in use of mobile mindfulness apps, with rolling admission and ascending practice dose ladder.
  2. MTPC (Mindfulness Training for Primary Care): An eight-week intensive mindfulness group with ascending practice dose ladder and skill integration over 8 weeks & 120 minutes/wk.
  3. MCS (Mindfulness Maintenance Check-in Support): Ongoing weekly mindfulness group with check-in and reminders, leveraging mobile mindfulness apps and motivational counseling for grads of LDM for 50 mins/wk.
  After completion of the LDM group, participation in various levels is fluid based on patient motivation, choice, and readiness.

SUMMARY:
The goal of this pilot study is to test the Mindful Recovery OBOT Care Continuum (M-ROCC) model in primary care office-based opioid treatment (OBOT). M-ROCC features integration of evidence-based mindfulness training with weekly group-based opioid treatment. Primary outcomes include (1) Feasibility measured by implementation of the curriculum into two CHA primary care sites and attendance at weekly sessions; (2) Acceptance via self-report and qualitative interviews. Secondary outcomes include anxiety reduction.

DETAILED DESCRIPTION:
The primary objective of this study is to conduct a single-arm pilot study in order to refine a Mindfulness-Based Intervention for the Opioid Use Disorder (OUD) treatment in primary care, called the Mindful Recovery OUD Care Continuum (M-ROCC). Study investigators will conduct qualitative interviews, assess opioid use, preliminary pre/post measures for participants participating in the pilot study. Additional aims of the pilot study is manual refinement and pilot testing assessment batteries to prepare for a multi-site RCT.

The study will focus on demonstrating feasibility and acceptability of the M-ROCC continuum.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Current CHA patient with a CHA primary care provider
3. Diagnosis of opioid use disorder prescribed buprenorphine/naloxone
4. Sufficient English fluency to understand procedures and questionnaires
5. <90 days of complete abstinence from illicit opioids, cocaine, benzodiazepines, AND alcohol (excluding cannabis/nicotine)
6. Ability to provide informed consent.

Exclusion Criteria:

1. Psychosis
2. Mania
3. Thought disorder
4. Schizophrenia or Schizoaffective disorder
5. Acute suicidality with plan
6. Cognitive inability as demonstrated by Montreal Cognitive Assessment (MOCA) <24 OR the inability to complete consent quiz and baseline assessments.
7. Current participation in another CHA research study
8. Expected hospitalization in next 6 months, including second and third trimester pregnancy at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Likelihood of recommending program to a friend | Week 24
  Percentage of participants who would recommend the program to a friend (score of 4 or 5 on a Likert scale (1-5))

SECONDARY OUTCOMES:
Number of weekly sessions attended | Week 24
  Percentage of attendance out of 24 weekly group sessions during the 6 month study period.
Anxiety PROMIS-SF 8a | Week 24
  The Patient Reported Outcomes Measurement Information System - Anxiety Short Form 8a (PROMIS-ASF) is an 8-item scale used to assess patient-reported health status for anxiety. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Subjects are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always). With use of the PROMIS Assessment Center Scoring Service, a T score is generated from subject responses. A sample item includes "My worries overwhelmed me."
Number of biochemically-confirmed illicit opioid abstinent weeks | Week 24
  Number of 2-week time periods with no self-reported illicit opioid use and biochemically-confirmed abstinence from illicit opioid use during a 24-week period. Urine toxicology will be administered every two weeks for 24 weeks and weekly self-report about illicit opioid use will be collected weekly.
PROMIS-SF 8a (PROMIS-ASF) Pain Interference | Week 24
  The PROMIS Pain Interference instruments measure the self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Pain Interference also incorporates items probing sleep and enjoyment in life, though the item bank only contains one sleep item. The Pain Interference short form is universal rather than disease-specific. It assesses pain interference over the past seven days. each question has five response options ranging in value from one to five (for pediatrics and parent proxy it is 0 to 4). To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 6-item form, the lowest possible raw score is 6; the highest possible raw score is 30. A higher PROMIS T-score represents higher consequences of pain.

OTHER OUTCOMES:
Number of biochemically-confirmed cocaine abstinent weeks | Week 24
  Number of 2-week time periods with no self-reported cocaine use and biochemically-confirmed abstinence from cocaine use during a 24-week period.
Brief Experiential Avoidance Questionnaire (BEAQ) | Week 24
  The Brief Experiential Avoidance Questionnaire (BEAQ) is a 15-item scale developed to assess a broad range of experiential avoidance (EA) content. Answers are based on a 6-point Likert scale. Total score is sum of individual items (range is 15 - 90). Higher score indicates higher levels of experiential avoidance.
Patient Reported Outcomes Measurement Information System - Depression Short Form (PROMIS-DSF) | Week 24
  The Patient Reported Outcomes Measurement Information System - Depression Short Form 8a (PROMIS-DSF) is an 8-item scale used to assess patient-reported health status for depression. PROMIS instruments are funded by the National Institutes of Health (NIH) and used to reliably and validly measure patient-reported outcomes for clinical research and practice. Participants are asked to rate their experience of the item in the past seven days on a 5-point scale from 1 (Never) to 5 (Always).
Five Facet Mindfulness Questionnaire (FFMQ) | Week 24
  is a 39-item scale that examines five factors that represent aspects of the current empirical conception of mindfulness. These five facets include: "observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience." An example item is "I pay attention to how my emotions affect my thoughts and behavior." Subjects rate their degree of agreement with each of the items on a Likert-type scale ranging from 1 (Never or very rarely true) to 5 (Very often or always true), with higher scores indicating higher experience of mindfulness. Total score is sum of all facets (range is 39 - 195). Subscales range from 7 - 40.
Difficulties in Emotion Regulation (DERS) Scale | Week 24
  The DERS is a 36-item self-report scale designed to assess emotional dysregulation. The scale assess 6 aspects of emotional dysregulation: non-acceptance of emotional responses ("When I'm upset, I become embarrassed for feeling that way"), difficulties engaging in goal directed behavior ("When I'm upset, I have difficulty thinking about anything else"), impulse control difficulties ("When I'm upset, I lose control over my behaviors"), lack of emotional awareness ("When I'm upset, I take time to figure out what I'm really feeling (reverse-scored)", limited access to emotion regulation strategies ("When I'm upset, it takes me a long time to feel better"), and lack of emotional clarity ("I have no idea how I am feeling"). Answers are selected from a 1-5 Likert scale. Total score is sum of each subscale. Subscales are scored by summing individual subscale items. Total score ranges from 36 to 180 and subscale scores range from 5 to 40.
Perceived Stress Scale (PSS) Scale | Week 24
  The PSS Scale uses 14 items to measure the degree to which situations in life are stressful. Items are designed to evaluate how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5 point Likert scale from 0 (Never) to 4 (Very often). An example question is, "In the last month, how often have you felt difficulties were piling up so high that you could not overcome them?" Positively stated items are reverse scored before all scale items are summed to yield a total score. Total score ranges from 0 to 56.
Self-Compassion Scale-Short Form (SCS-SF) | Week 24
  The short-form Self-Compassion Scale (SCS-SF) is an abbreviated 12-item form of the original 26-item Self-Compassion Scale. The scale is scored on a 5 point Likert scale (1 = Almost never; 5 = Almost always), and negative subscale items are reverse scored. Total score is calculated by taking the mean of all scores and ranges from 1 to 5.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Week 24
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item self-report scale designed to assess multiple aspects of interoception and interoceptive awareness. The 6 point Likert scale (ranging from 0-5) assesses 8 aspects of interoceptive awareness: noticing, not-distracting, not-worrying, attention regulation, emotional awareness, self-regulation, body listening, and trusting. Subscales are averaged, and a higher total score represents a better outcome. Total average score can also be reported. Total and subscale scores range from 0 to 5.
Sustained Attention to Response Task (SART) | Week 24
  Participants complete a computerized test measuring sustained attention and response inhibition. They are asked to press a key in response to rapidly displayed integers (1-9) and withhold a response to a designated "no-go" integer.
Hypothetical Delay Discounting Task (HDT) | Week 24
  This is a brief delay discounting task performed on a computer that presents a series of 5 discrete choice questions between delayed larger reward and smaller sooner reward in dollars.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Cambridge Health Alliance, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fatkin T, Moore SK, Okst K, Creedon TB, Samawi F, Fredericksen AK, Roll D, Oxnard A, Le Cook B, Schuman-Olivier Z. Feasibility and acceptability of mindful recovery opioid use care continuum (M-ROCC): A concurrent mixed methods study. J Subst Abuse Treat. 2021 Nov;130:108415. doi: 10.1016/j.jsat.2021.108415. Epub 2021 Apr 15. PMID 34118705
- [Result] Schuman-Olivier Z, Fatkin T, Creedon TB, Samawi F, Moore SK, Okst K, Fredericksen AK, Oxnard AS, Roll D, Smith L, Cook BL, Weiss RD. Effects of a trauma-informed mindful recovery program on comorbid pain, anxiety, and substance use during primary care buprenorphine treatment: A proof-of-concept study. Am J Addict. 2023 May;32(3):244-253. doi: 10.1111/ajad.13364. Epub 2022 Dec 5. PMID 36470641

DOCUMENTS (1):
  • Informed Consent Form (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03798431/ICF_002.pdf